CLINICAL TRIAL: NCT02779231
Title: Hypertension Control Using Bi-directional Texting for Home Blood Pressure Monitoring
Brief Title: Text Messages and Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linnea Polgreen (Other)
Responsible Party: Sponsor-Investigator, Linnea Polgreen, M.D., University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201509761
Record Dates: First submitted 2016-05-16; First posted 2016-05-20 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Texting group (Experimental): This group will be enrolled in bi-directional texting to send back blood pressure.
  Interventions: Other: Bi-directional texting
- Standard of care group (No Intervention)

INTERVENTIONS:
Other: Bi-directional texting
  Arms: Texting group

SUMMARY:
Hypertension remains one of the most important preventable contributors to disease and death. It is the most common risk factor for strokes and myocardial infarctions in the U.S., and is associated with the greatest attributable risk for mortality among all modifiable risk factors for cardiovascular events. Over 50 million people are living with hypertension in the United States, and hypertension is one of the most common reasons for visits to a healthcare provider. Abundant evidence from randomized controlled trials has shown benefit of antihypertensive drug treatment in reducing important health outcomes in persons with hypertension. Yet, approximately 20% of U.S. adults are unaware that they have the disease.

Hypertension is more difficult to diagnose than other common medical illnesses. In most cases, hypertension is asymptomatic; and accordingly patients do not seek care for it as they do for other common symptomatic illness. Patients are frequently diagnosed after presenting with end organ disease (e.g., myocardial infarctions, congestive heart failure, strokes, or renal failure). Another complicating aspect related to diagnosing uncontrolled hypertension is that multiple blood pressure measurements are needed to establish a diagnosis. Blood pressure readings can be falsely elevated in clinic due to the presence of an observer or the clinical surrounding (e.g., white coat hypertension). Even if an elevated blood pressure reading is identified in a clinic setting, more readings are needed in order to make it possible for physicians to decide about the next appropriate medical intervention. This need for multiple BP measurements over time often delays both initiating and modifying medical therapy for uncontrolled hypertension.

Having patients take their BP at home facilitates the more timely diagnosis of uncontrolled hypertension by reducing diagnostic uncertainty. In fact, home measurements are better diagnostic indicators of stroke and cardiovascular mortality than clinic readings, are more closely correlated with end-organ damage, and are cost effective and well-tolerated by patients.

Patients are frequently asked to record their BP after clinic visits. Historically, patients used a hand-written log, but more recently, patients are instructed to use an Internet-based web portal that uploads values to the patient's electronic medical record. Compliance with either approach relies on effective patient and provider followup, and in many settings, nurses or pharmacists will need to call patients to prompt them for their blood pressure measurements, which is both a costly and time consuming approach. Therefore, researchers need to develop effective, yet low cost alternatives to monitoring home blood pressure.

This study proposes such a solution. The purpose of this study is to evaluate a simple m-health intervention to increase the ease and efficacy of diagnosing uncontrolled hypertension and achieve better blood pressure control in hypertensive patients.

DETAILED DESCRIPTION:
Half of the participants will be randomized to a "text-messaging" protocol, and the other half will be randomized to a "standard of care" protocol.

Text messaging protocol: A trained research personnel (student, pharmacist, physician or research assistant) will record the patient's cell phone number. Participants will select 7 morning and 7 evening times that are convenient for them to check and send blood pressure measurements. (The literature recommends that 12-14 measurements should be taken over one to weeks with morning and evening readings before making a diagnosis of hypertension). Participants will use a home blood pressure monitor that will be provided to them after given instruction of how to use it. This visit should take around 30 minutes.

After the participant leaves the clinic, at the pre-specified times and dates, an automated server side script running on the investigators' server will check the application database at a given time interval and at the appropriate times send the participant a text message with specific, simple instructions. An example of the message is as follows: "Please remember to check your blood pressure this morning at 7am! Reply to this message with your blood pressure and time it was taken." The participant will return a short text with his/her blood pressure measurements and the time they were taken: "150/90 and 145/88 7am". The investigators' software will identify the cell phone number associated with each message and will enter the blood pressure measurement, the time the blood pressure was recorded, and the time the message was received into an account associated with that participant in our secure database. If the participant does not complete the blood pressure homework assignment, a pre-specified number of reminders will be sent to the patient until 2 weeks have elapsed.

Once the pre-specified number of measurements (seven days' worth of measurements) has been received by the website, an email alert will be sent to the study personnel and a generated document with blood pressure numbers will be sent to the treating physician e.g. physician's clinical mailbox.

Standard of care protocol: participants who are randomized to the "Standard of Care" group will be instructed to obtain 7 morning and 7 evening blood pressure measurements. Participants will be asked to choose a method of communication to reply their blood pressure numbers back to their physician. These include "MyChart" which is Internet-based web-portal connected to the participant's electronic medical record, calling back the clinic with their numbers, mailing, or faxing blood pressure log to their physician. The type of method each participant chooses will be recorded. Participants will use a home blood pressure monitor that will be provided to them after given instruction on how to use it.

Participants in both groups will be asked to return the blood pressure cuff to Iowa River Landing Internal Medicine clinic. This can be done at any time that is convenient to them after finishing the blood pressure assignment.

During the study, investigators will access the participants' medical record to obtain the following information: latest blood pressure measurement, blood pressure medications, latest cholesterol measurements, cholesterol medications, latest glucose measurement, other chronic medical conditions, other medications, insurance, race, age, gender, marital status, height and weight.

Medical records will also be accessed 3-6 months later to identify any change in medical management that occurred after sending blood pressure readings. Time and type of intervention will be recorded whether it is adding a new medication or increasing a current medication dose. Also blood pressure readings during the next clinic visit (3-6 months after the study) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with at least one high blood pressure during any clinic visit over the past 6 months who owns cell phone with texting capability.
* Eligible participants will be asked the following screening questions:

  * "Do you have a cell phone with text messaging ability?", and "are you willing to send your blood pressure numbers through text messages?". The participant should answer "yes" to both questions to be eligible for the study.

Exclusion Criteria:

* Active or acute mental health problem;
* Significant cognitive impairment;
* Lack of fluency in speaking or understanding English;
* Pregnancy.
* Also, If the participant answers "NO" to any one of the screening two questions, they will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Patients' response to texting. | 15 days
  The number of participants who completed the home blood pressure assignment will be compared between the two groups. These data will be extracted from the medical records for the standard of care group and from the "texting" website for the texting group.
Physicians' response to blood pressure information. | 30 days
  The number of physicians who reacted to the blood pressure readings with any kind of clinical intervention (life style discussion, medication modification, ets.) will be compared between the two groups. These data will be extracted from the medical records.
Diagnosis rates between the text-messages and the standard of care groups. | 6 months

SECONDARY OUTCOMES:
Time to intervention by physicians between the two groups | 30 days
Difference in blood pressure reduction between the two groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip Polgreen, M.D. Ph.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States